CLINICAL TRIAL: NCT02468388
Title: Study on the Effect of Chewing Sugar-free Gum on Re-mineralization of Early Caries Via Quantitative Light-induced Fluorescence
Brief Title: Re-mineralization Effects of Sugar Free Chewing Gum Sweetened With Different Sugar-substitutes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roquette Management (Shanghai) Co., Ltd. (Industry)
Collaborators: West China College of Stomatology (Other); Kaunas University of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CPS 10-341
Record Dates: First submitted 2015-06-03; First posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Re-mineralization
Keywords: maltitol; xylitol; quantitative light-induced fluorescence; saliva pH; re-mineralization; dental caries
MeSH Terms: conditions — Dental Caries | interventions — maltitol; Xylitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- maltitol (Experimental)
  Interventions: Other: maltitol
- xylitol (Active Comparator)
  Interventions: Other: xylitol
- gum base (Placebo Comparator)
  Interventions: Other: gum base
- no gum (No Intervention)

INTERVENTIONS:
Other: maltitol — maltitol chewing gum: 66% SweetPearlTM Maltitol +30.91% gum base+1.93% Lycasin R 85/55+0.39% glycerin; two pellets for 10 min five times each day
  Arms: maltitol
Other: xylitol — xylitol chewing gum: 67.73% xylitol +30.02% gum base+1.13% Lycasin R 85/55+0.38% glycerin; two pellets for 10 min five times each day
  Arms: xylitol
Other: gum base — gum base: 99% gum base; two pellets for 10 min five times each day
  Arms: gum base

SUMMARY:
The purpose of this study is to evaluate the clinical effect of chewing gum containing maltitol, on re-mineralization of early caries following daily chewing for 6 months by school children, compared to a xylitol gum, gum base and a no gum group.

ELIGIBILITY:
Inclusion Criteria:

* Consent Informed Consent Form signed by parent or legal guardian permitting participation of their children.
* Be cooperative and able to be examined in the whole study duration.
* Aged from 8 to 13 years.
* General Health: Good general health (in the opinion of the investigator) without clinically significant and relevant abnormalities of medical history such as diabetic, etc.
* Oral Health: Display 6 permanent front teeth and two maxillary buccal surfaces with visual evidence of active initial enamel carious lesions (de-mineralized but not cavitated); No any form of intraoral prostheses or appliances, clinical signs of severe gingivitis or periodontitis, temporomandibular joint disorders, and malocclusions or chronic onychophagia
* Oral Hygiene: have good oral health habits, brushing teeth at least once per day
* No medical or pharmacotherapy history that might affect the outcomes of the study, e.g. use of mouthwash, gels, or chewing gum containing antimicrobial agents during the previous 3 months

Exclusion Criteria:

* Disease: Presence of chronic debilitating disease, or any condition or other chronic disease which the investigators think not suitable for the study.
* Allergy/Intolerance: Be allergic to both maltitol and xylitol, oral care products, personal care consumer products, or their ingredients.
* Current Product Use: usual chewing-gum (of any kind) consumer or sugars-free candies consumer
* Clinical Study/Experiment: Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 482 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in re-mineralization of early caries at 3 months measured by quantitative light-induced fluorescence | baseline and 3 months
Change from baseline in re-mineralization of early caries at 6 months measured by quantitative light-induced fluorescence | baseline and 6 months

SECONDARY OUTCOMES:
Change from baseline in Streptococcus mutans counts in saliva at 3 months measured by Dentocult strip | baseline and 3 months
Change from baseline in Streptococcus mutans counts in saliva at 6 months measured by Dentocult strip | baseline and 6 months
Change from baseline in Potential hydrogen (pH) of saliva at 3 months measured by pH meter | baseline and 3 months
Change from baseline in Potential hydrogen (pH) of saliva at 6 months measured by pH meter | baseline and 6 months
Change from baseline in Silness & Loe Plaque index at 3 months | baseline and 3 months
Change from baseline in Silness & Loe Plaque index at 6 months | baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Deyu Hu, Ph.D., Principal Investigator — West China College of Stomatology, Sichuan University
Locations (1):
- West China College of Stomatology, Sichuan University, Sichuan, Sichuan, China